CLINICAL TRIAL: NCT04319068
Title: Sodium Storage in Singaporeans
Acronym: SSIS
Status: Active, not recruiting | Type: Observational
Sponsor: Jens Titze (Other)
Collaborators: National Heart Centre Singapore (Other)
Responsible Party: Sponsor-Investigator, Jens Titze, Associate Professor, Duke-NUS Graduate Medical School
Organization: Duke-NUS Graduate Medical School (Other)
Other Study IDs: SSIS
Record Dates: First submitted 2020-03-18; First posted 2020-03-24 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Healthy; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine and Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy: Eligible participants from the Biobank cohort at the National Heart Centre, Singapore, will be screened will be recruited for the study over a period of 3 years.
- Hypertensive: Eligible participants from the Biobank cohort at the National Heart Centre, Singapore, will be screened will be recruited for the study over a period of 3 years

SUMMARY:
The overarching hypothesis of this study is that the kidney and the skin form an integrative network for water conservation, where Na+ storage is utilized to prevent body water loss, even at the expense of increased cardiovascular risk. The aim of this project is to characterise skin and muscle Na+ storage in a cohort designed to prospectively measure cardiovascular outcomes in Singaporeans, in order to determine whether humans with increased tissue Na+ storage have increased cardiovascular risk. To gain a better understanding of the mechanisms behind Na+ storage, the investigators will also test the hypothesis that participants with mutations of the skin protein filaggrin, who have increased water loss through the skin, will have increased skin Na+ storage and higher blood pressure levels.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) occurs with increasing age and is the leading cause of death worldwide. A causal relationship between salt and CVD, although well established in animal models, has been difficult to prove in human populations. First, because humans do not live under the strict experimental conditions necessary to quantify sodium intake, and second, because tissue sodium stores cannot be detected with the available clinical methods, making reliable measurements of total body sodium extremely challenging.

The investigators have previously implemented 23NaMRI technology to detect and quantify tissue Na+ stores in humans. Previous studies have sown that humans store large amounts of Na+ in their skin and muscle as they age and that skin Na+ storage is linked with hypertension, while muscle Na+ storage is coupled with insulin resistance and diabetes. More recent studies show that the adverse effect of Na+ on human health goes far beyond the well-established salt-blood pressure relationship. The investigators have found that urea and/or Na+ storage in barriers such as kidney or skin is a key principle of water conservation.

This study aims to test the hypothesis that water conservation in the skin is essential for systemic fluid and blood pressure homeostasis, and that skin Na+ storage is utilized to prevent water loss, even at the expense of increased cardiovascular risk.

This is a cross-sectional study design with one study visit and a recruitment period of 3 years. 600 participants will be recruited from the Biobank cohort and tissue Na+ will be measured using 23NaMRI. The study will test whether increased Na+ storage in the skin is coupled with transepidermal water loss at the expense of high blood pressure levels, and examine the association between tissue sodium storage and specific cardiovascular markers.

ELIGIBILITY:
Inclusion Criteria:

1. Participants from the Biobank (Molecular and Imaging Studies of Cardiovascular Health and Disease) cohort in Singapore, who agreed to be contacted for further studies
2. Male and female patients older than 21 years
3. Willingness to participate and ability to provide informed consent

Exclusion Criteria:

1. Patients with exclusion criteria for the MRI, such as:

   1. implanted devices (surgical clips, heart pacemakers or defibrillators, cochlear implants)
   2. iron-based tattoos
   3. any other pieces of metal or devices that are not MR-Safe anywhere in the body
   4. patients who exhibit noticeable anxiety and/or claustrophobia into the MRI scanner
2. Pregnant women
3. Diagnosis of heart failure NYHA classes III and IV
4. Impaired renal function with eGFR<45 ml/min or proteinuria > 0.5 g/24h
5. Liver disease with cirrhosis (Child-Pugh class C) or hypoalbuminemia
6. Peripheral oedema as assessed by the investigator
7. Active cancer
8. Patients who have received an organ or bone marrow transplant
9. Patients who have had major surgery in the past 3 months
10. Patients who have severe comorbid conditions likely to compromise survival or study participation
11. Unwillingness or other inability to cooperate

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible participants from the Biobank cohort at the National Heart Centre, Singapore, will be screened and estimated 600 subjects (healthy controls and hypertensive patients) will be recruited for the study over a period of 3 years. No ethnic group or gender is targeted for or excluded from this reasearch.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-07-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Skin and muscle Na+ content | 3 years
  Differences in skin and muscle Na+ content (measured with 23NaMRI) between healthy participants and hypertensive patients, overall and according to age, gender and race/ethnicity

SECONDARY OUTCOMES:
Correlation between skin water loss and skin Na+ content | 3 years
  To show that participants with high transepidermal water loss (measured with Tewameter TM300) have higher skin sodium content (measured with 23NaMRI)
Skin water loss in hypertensive participants | 3 years
  To show that hypertensive participants have higher transepidermal water loss (measured with Tewameter TM300) and higher skin Na+ content than healthy participants

CONTACTS AND LOCATIONS:
Locations (2):
- Singapore (2):
  - National Heart Centre Singapore, Singapore
  - Duke-NUS Medical School, Singapore

REFERENCES:
- [Background] Kopp C, Linz P, Dahlmann A, Hammon M, Jantsch J, Muller DN, Schmieder RE, Cavallaro A, Eckardt KU, Uder M, Luft FC, Titze J. 23Na magnetic resonance imaging-determined tissue sodium in healthy subjects and hypertensive patients. Hypertension. 2013 Mar;61(3):635-40. doi: 10.1161/HYPERTENSIONAHA.111.00566. Epub 2013 Jan 21. PMID 23339169
- [Background] Titze J. Sodium balance is not just a renal affair. Curr Opin Nephrol Hypertens. 2014 Mar;23(2):101-5. doi: 10.1097/01.mnh.0000441151.55320.c3. PMID 24401786
- [Background] Schneider MP, Raff U, Kopp C, Scheppach JB, Toncar S, Wanner C, Schlieper G, Saritas T, Floege J, Schmid M, Birukov A, Dahlmann A, Linz P, Janka R, Uder M, Schmieder RE, Titze JM, Eckardt KU. Skin Sodium Concentration Correlates with Left Ventricular Hypertrophy in CKD. J Am Soc Nephrol. 2017 Jun;28(6):1867-1876. doi: 10.1681/ASN.2016060662. Epub 2017 Feb 2. PMID 28154199
- [Background] Titze J. Estimating salt intake in humans: not so easy! Am J Clin Nutr. 2017 Jun;105(6):1253-1254. doi: 10.3945/ajcn.117.158147. Epub 2017 May 17. No abstract available. PMID 28515066
- [Background] Rakova N, Kitada K, Lerchl K, Dahlmann A, Birukov A, Daub S, Kopp C, Pedchenko T, Zhang Y, Beck L, Johannes B, Marton A, Muller DN, Rauh M, Luft FC, Titze J. Increased salt consumption induces body water conservation and decreases fluid intake. J Clin Invest. 2017 May 1;127(5):1932-1943. doi: 10.1172/JCI88530. Epub 2017 Apr 17. PMID 28414302